CLINICAL TRIAL: NCT01947049
Title: Influenza Diagnosis, Treatment and Surveillance With Xpert Flu
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Principal Investigator, Rich Rothman, Professor, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 6 IDSEP130014-01-01
Record Dates: First submitted 2013-09-17; First posted 2013-09-20 (Estimated); Last update posted 2017-09-18 (Actual); Status verified 2017-09

CONDITIONS: Influenza
Keywords: Influenza; diagnostic testing; antiviral treatment; rapid influenza testing
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Arm (No Intervention): Participants in this arm will receive usual care (influenza testing and treatment)
- Rapid Testing (Experimental): Participants in this arm will receive rapid influenza testing with Xpert Flu.
  Interventions: Other: Rapid Influenza Testing with Xpert Flu

INTERVENTIONS:
Other: Rapid Influenza Testing with Xpert Flu — Participants with recieve rapid influenza testing with Xpert Flu
  Arms: Rapid Testing

SUMMARY:
The purpose of this study is to:

1. Evaluate the clinical performance of a newly available highly-sensitive rapid influenza test, Xpert Flu.
2. Derive and validate an adult clinical decision guideline to guide clinical testing of influenza patients who meed CDC criteria for antiviral treatment.
3. Evaluate impact of rapid influenza testing for antiviral treatment.
4. Determine cost effectiveness of influenza testing and treatment strategies.

DETAILED DESCRIPTION:
Four strategically selected medical centers across the US (representing the West Coast, Southwest, Midwest; and East Coast) will enroll adult subjects presenting to the ED with an acute respiratory illness who fulfill CDC recommended criteria for receiving antiviral therapy. At each of the 4 sites, dedicated research coordinators will approach all adult (age > 18 years old) ED patients with broadly defined respiratory related complaints and screen for those who meet CDC recommended criteria for antiviral therapy (i.e. those at 'high-risk for complications' or those with 'potential influenza-related complications).

Consenting subjects will have a nasopharyngeal (NP) swab collected for both Xpert Flu testing and gold standard reverse transcription-PCR (rt-PCR) testing under a research protocol. The investigators will compare the test results from the rapid flu testing to that of the gold standard rt-PCR testing in order to assess the clinical performance characteristics of the new rapid test (Objective 1). The investigators will also collect demographics and medical historical information using a brief structured data form, which will be used in combination with rt-PCR test results to derive and validate a clinical decision guideline (Objective 2).

The investigators will simultaneously randomize 2 of the 4 hospitals to the Rapid Testing Group (which will have systematic rapid flu testing performed with results provided to the clinicians), or the Control Group (which will follow standard of care practice with testing left to the discretion of individual clinicians). This will permit comparison of rates of ED antiviral administration or prescription between the two groups to assess the clinical impact of influenza testing (Objective 3). Finally, cost data from the ED visits and subsequent hospitalization will be collected from subjects in both the rapid testing group and the control group to inform a cost-utility analysis of rapid influenza testing compared to current standard of care (Objective 4).

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* Acute respiratory tract infection, i.e. in the past two days the subject has experienced any of the following symptoms: new or increased cough, new or increased shortness of breath, change in sputum production (for adults 65 years or older), new sinus pain, new nasal congestion/rhinorrhea, new sore throat, new fever, triage temperature greater than or equal to 38F
* CDC Criteria for influenza antiviral treatment, i.e. is the subject at risk for influenza complications or does the subject have potential current influenza complications including: 65 years old or older, pregnant (or less than 2 weeks post-partum), American Indian or Alaska Native, morbid obesity (BMI greater than 40), current resident of a chronic care facility, chronic pulmonary disease, cardiovascular disease (except isolated hypertension), renal disease, hepatic disease, hematologic disease, metabolic disease, neurologic disease, immunosupression due to [HIV or AIDS, transplant, chemotherapy, medications, other - specify]. OR does the subject have potential current influenza complications such as: admitted to the hospital or a diagnosis of pneumonia.

Exclusion Criteria:

* Unable to speak or understand English or Spanish
* Unable to provide consent
* Lack of follow up information (i.e. working telephone number)
* Have an influenza diagnosis in the past 2 weeks (i.e. either given antivirals or had a confirmatory influenza test)
* Previously enrolled in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2011 (Actual)
Dates: Start 2013-07; Primary Completion 2014-06-30 (Actual); Study Completion 2014-06-30 (Actual)

PRIMARY OUTCOMES:
Clinical performance of Xpert Flu | one year
  The primary outcome is the sensitivity and specificity of Cepheid Xpert Flu in detecting Influenza, as well as the positive and negative predictive value.

SECONDARY OUTCOMES:
Clinical decision guideline | one year
  Using rt-PCR as the gold standard for influenza testing, we will initially evaluate signs and symptoms (such as cough, fever, sore throat, shortness of breath, etc.) for their sensitivity, specificity and likelihood ratio for diagnosing influenza.
Clinical Utility of Xpert Flu | one year
  Clinical utility is defined here as the proportion of high-risk subjects with confirmed influenza receiving antiviral or antiviral prescriptions in the ED in the Rapid Testing Group compared to the Control Group.
Cost-effectiveness | one year
  We will perform a cost-utility analysis from the societal perspective comparing the following 4 treatment strategies: 1) treat all; 2) treat none; 3) treat based on clinical judgment; 4) treat based on Xpert Flu.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Dugas, MD, Principal Investigator — Johns Hopkins University; Richard Rothman, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (4):
- United States (4):
  - Maricopa Medical Center, Phoenix, Arizona
  - Olive View - UCLA Medical Center, Sylmar, California
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Truman Medical Center, Kansas City, Missouri

REFERENCES:
- [Derived] Dugas AF, Hsieh YH, LoVecchio F, Moran GJ, Steele MT, Talan DA, Rothman RE; Emergency Department National Influenza Network Investigators. Derivation and Validation of a Clinical Decision Guideline for Influenza Testing in 4 US Emergency Departments. Clin Infect Dis. 2020 Jan 1;70(1):49-58. doi: 10.1093/cid/ciz171. PMID 30843056